CLINICAL TRIAL: NCT01267617
Title: Measuring Cardiovascular Stress in Patients on Hemodialysis
Status: Completed | Type: Observational
Sponsor: West Penn Allegheny Health System (Other)
Responsible Party: Rita L. McGill MD, West Penn Allegheny Health System
Other Study IDs: RC-5046
Record Dates: First submitted 2010-12-23; First posted 2010-12-28 (Estimated); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Hemodialysis; Hypotension; Circulatory Stress; Photo-plethysmography
Keywords: hemodialysis; hypotension; circulatory stress; photo-plethysmography
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- chronic hemodialysis outpatients

SUMMARY:
To determine if proprietary software that uses pulse-wave analysis to interpret the output of a conventional pulse-oximeter, can predict the onset of circulatory stress, before changes in blood pressure and pulse occur, in patients undergoing outpatient hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients having regular outpatient dialysis treatments
* Patients who are willing and able to provide informed consent

Exclusion Criteria:

* Patients who do not wish to participate
* Patients with contraindications to attachment of monitoring devices
* Patients with skin rash or hypersensitivity to the adhesive sensors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients receiving hemodialysis at a single center
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2010-11-30 (Actual); Primary Completion 2011-11-14 (Actual); Study Completion 2011-11-14 (Actual)

PRIMARY OUTCOMES:
photoplethysmography | 5 hours
  Pulse-wave analysis of an oximeter signal

SECONDARY OUTCOMES:
blood pressure | 5 hours
  measured continuously during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Rita L McGill, MD, Principal Investigator — West Penn Allegheny Health System
Locations (1):
- Allegheny General Hospital, Pittsburgh, Pennsylvania, United States